CLINICAL TRIAL: NCT03378960
Title: Bioavailability Study of Omeprazole (20 mg) at Steady State (Multiple Dose) in Patients Who Have Undergone Bariatric Surgery
Brief Title: Study to Compare the Bioavailability of Omeprazole 20 mg Before and After Undergoing Surgery for Morbid Obesity
Acronym: OBS-2011/001
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emilio Vargas Castrillón (Other)
Collaborators: Fundación Mutua Madrileña (Other)
Responsible Party: Sponsor-Investigator, Emilio Vargas Castrillón, Head of Clinical Pharmacology Department, Hospital San Carlos, Madrid
Organization: Hospital San Carlos, Madrid (Other)
Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: OBS-2011/001
Record Dates: First submitted 2017-11-27; First posted 2017-12-20 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Bariatric Surgery Candidate
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Intervention Model Description: This was a single-dose, open-label, bioavailability study of surgical group and controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- omeprazole (Other): omeprazole 20 mg
  Interventions: Drug: Omeprazole 20mg

INTERVENTIONS:
Drug: Omeprazole 20mg

SUMMARY:
The principal aim was to evaluate whether gastric bypass surgery modifies the bioavailability of omeprazole 20 mg at one month and six months after surgery.

Other objectives were:

* To compare bioavailability of omeprazole 20 mg between patients undergo gastric bypass surgery and patients who avoid it.
* To asses other pharmacokinetic parameters, demographic parameters and drug safety.

Study design It was planned a mixed design which intended to compare the bioavailability in patients with gastric bypass (before and after surgery) and control subjects matched by sex and body mass index (BMI) post-surgery. This was a single-dose, open-label, crossover bioavailability study of omeprazole in surgical group and controls.

ELIGIBILITY:
Inclusion Criteria:

* Patients who wish to participate in the study (men and women) after receiving adequate information about the study design, objectives and risks by signing and date of the written informed consent.
* Age between 18 and 60 years old.
* Patients who come to the endocrinology and nutrition Service and on treatment with omeprazole.
* Patients who are to undergo bariatric surgery (Roux en Y gastric bypass) according to the recommendations of Endocrinology and Nutrition Service and the Department of General Surgery and Digestive Diseases hospital Clinico San Carlos.
* No significant abnormalities on clinical examination and laboratory analysis before inclusion in the study.

Exclusion Criteria:

* Any postoperative complication that interferes with the regular intake of medication such as stenosis of anastomotic, fistula, persistent vomiting, diarrhea (> 4 stools per day), evidence of protein malnutrition (albumin <3.5 g / l).
* High consumption of stimulating beverages (equivalent to 400 mg of caffeine per day, a cup of coffee contains approximately 100 mg of caffeine).
* Consumption of any medication that may interfere with the objectives of the study: * Use of enzyme inhibitors or inducers within 2 weeks prior to study inclusion (barbiturates, carbamazepine, erythromycin, phenytoin, oral contraceptives, etc.) * Any concomitant medication will be assessed by the investigator based on data recorded in the log-book for the medication (potential interactions) and registered in the CRF.
* History of clinically significant disease in the opinion of the investigator does not allow safe participation of the patient.
* Inability to relate to and / or cooperate with investigators.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2014-10-31 (Actual); Primary Completion 2015-12-23 (Actual); Study Completion 2016-02-29 (Actual)

PRIMARY OUTCOMES:
AUC variation Pharmacokinetic parameters | Baseline and 6 month after bariatric surgery
  Omeprazole Biodisponibility
Tmax variation | Baseline and 6 month after bariatric surgery
  Time required to reach the maximum concentration of Omeprazole in blood after its administration.
Cmax variation | Baseline and 6 month after bariatric surgery
  Maximum concentration of Omeprazole in blood after its administration.

SECONDARY OUTCOMES:
AUC 1 month | 1 month after surgery
  Omeprazole Biodisponibility
Tmax 1 month | 1 month after surgery
  Time required to reach the maximum concentration of Omeprazole in blood after its administration
Cmax 1 month | 1 month after surgery
  Maximum concentration of Omeprazole in blood after its administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundacion para Investigación Biomedica Hospital Clinico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No